CLINICAL TRIAL: NCT05353504
Title: "SFB 1052/3 - Mechanismen Der Adipositas, Projekt A1: Veränderung Der Neurobiologischen Grundlagen Von Ess-Entscheidungen Bei Adipositas" Engl. "CRC 1052/3 - Obesity Mechanisms, Project A1: Targeting Neurobehavioral Determinants of Obesity"
Brief Title: Impact of Microbiome-changing Interventions on Food Decision-making
Acronym: MIFOOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Collaborators: Universitätsklinikum Leipzig (Other); DFG - Deutsche Forschungs Gemeinschaft (German Research Foundation) (Unknown); Helmholtz-Zentrum für Umweltforschung - UFZ (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MIFOOD
Record Dates: First submitted 2022-03-23; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: People will be randomly assigned to the three arms and blinded towards receipt of dietary fibre supplement or placebo supplement. However, behavioural lifestyle intervention arm cannot be blinded to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- prebiotic dietary supplement (Active Comparator): high-dose daily inulin
  Interventions: Dietary Supplement: Inulin
- behavioural lifestyle intervention (Experimental): new educational program to change eating behaviour, provided through weekly sessions.
  Interventions: Behavioral: Lifestyle intervention
- placebo dietary supplement (Placebo Comparator): equicaloric daily maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin — 28g/day delivered in 2 sachets throughout the day with main meals
  Arms: prebiotic dietary supplement
Behavioral: Lifestyle intervention — weekly educational sessions to improve individual's eating behaviour
  Arms: behavioural lifestyle intervention
Dietary Supplement: Placebo — equicaloric maltodextrin delivered in 2 sachets throughout the day with main meals
  Arms: placebo dietary supplement

SUMMARY:
The investigators aim to test the hypothesis that a microbiome-changing dietary intervention improves food decision-making and to determine the underlying microbiotal and metabolic mechanisms. To this end, 90 overweight/obese adults will be enrolled in a randomized controlled trial to test the effects of a pre-biotic dietary intervention (supplementary intake of soluble fibre) or a behavioural lifestyle intervention (weekly educational program) vs. control condititon (supplementary intake of isocaloric starch) over a period of 26 weeks. Before and after the intervention/control period, participants will undergo task-based functional and structural MRI and cognitive testing. The gut microbiota will be assessed using 16S rDNA next-generation sequencing (V3/V4 region) in stool samples. Diet, anthropometry and lifestyle will be monitored with questionnaires and metabolomics will be assayed in peripheral blood and stool (e.g. SCFA). Using a modulation of gut-brain communication through a prebiotic diet and lifestyle intervention, respectively, the investigators will be able to discover microbiota communities that play a key role for eating behaviour. Related mechanistic insights could help to develop novel preventive and therapeutic options to combat unhealthy weight gain in our obesogenic society.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 25 kg/m2 or WHR >= 0.9/0.85 (m/d, f)
* no MRI contra-indication
* written informed consent

Exclusion Criteria:

* athletes
* occurrence of a clinically relevant psychiatric disease in the last 12 months, e.g. depression, substance abuse, eating disorders, schizophrenia
* any chronic inflammatory or malignant disease
* type 1 diabetes
* previous bariatric/gastric surgery
* pregnancy or breastfeeding woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — all genders, self-report
Enrollment: 90 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
blood-oxygenation-level-dependent (BOLD) activity during food wanting | 6 months
  BOLD-acitvity will be measured using event-related echo-planar T2*-weighted magnetic resonance imaging (MRI) during food wanting task according to previously described procedures (details of preprocessing at: https://osf.io/ynkxw). Onsets of food and art stimuli presentation will be modelled as separate regressors convolving delta functions with a canonical hemodynamic response function. Wanting rating scores (on an 8-point likert scale) per stimulus will be added as covariates. In a parallel model, kcal of food stimuli will be added multiplied with wanting scores to model high caloric food wanting interaction. At the group level, we will assess the contrasts food > art and wanting modulation.

SECONDARY OUTCOMES:
microbial alpha and beta diversity | 6 months
  Changes in alpha and beta diversity assessed using 16S rRNA sequencing of stool samples
fMRI BOLD activity memory performance | 6 months
  BOLD-acitvity will be measured using event-related echo-planar T2*-weighted magnetic resonance imaging (MRI) during food wanting and food memory recognition tasks according to previously described procedures (details of preprocessing at: https://osf.io/ynkxw). Onsets of food and art stimuli presentation in encoding and recognition will be modelled as separate regressors convolving delta functions with a canonical hemodynamic response function. Correctly remembered and correctly rejected, as well as misses and false alarms will be modeled separately. In parallel models, similar and new items als well as wanting rating scores (on an 8-point likert scale) per stimulus and kcal of food stimuli multiplied with wanting scores will be added as covariates. At the group level, we will assess the contrasts correct > false and wanting modulation.
satiety | 6 months
  self-reported hunger feeling on a 8-point score from minimum 0 (not at all) to maximum 8 (very much).
ghrelin | 6 months
  ghrelin pg/ml in blood
leptin | 6 months
  leptin ng/ml in blood
GLP-1 | 6 months
  Glucagon-like peptide-1 (GLP-1) pg/ml in blood
PYY | 6 months
  peptide YY pg/ml in blood
insulin | 6 months
  insulin in blood uU/ml
HbA1c | 6 months
  hemoglycated globulin A1c in blood %
inflammatory markers | 6 months
  high sensitive C-reactive protein mg/l (and optionally tumor necrosis factor alpha and interleukin 6 in blood, pg/ml)
microbial metabolic markers in blood | 6 months
  short-chain fatty acids (SCFA), bile acids
body mass index | 6 months
  weight kg/height in m squared
waist hip ratio | 6 months
  waist (cm) to hip (cm) circumeference ratio
body fat | 6 months
  body fat % according to bioelectrical impedance analysis
food craving | 6 months
  assessed with the food craving questionnaire (Meule et al., 2012, German version).
executive attention performance | 6 months
  measured using the attention network task (ANT)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Witte, PhD, Principal Investigator — Cognitive Neurology, University Medical Center Leipzig
Locations (1):
- Department of Neurology, Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all data openly but anonymized on secured German servers of the institute after registration with ID.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: after end of study for 5 years or longer
Access Criteria: Registration on a website, providing copy of ID

REFERENCES:
- [Derived] Vartanian M, Endres KJ, Lee YT, Friedrich S, Meemken MT, Schamarek I, Rohde-Zimmermann K, Schurfeld R, Eisenberg L, Hilbert A, Beyer F, Stumvoll M, Sacher J, Villringer A, Christensen JF, Witte AV. Investigating the impact of microbiome-changing interventions on food decision-making: MIFOOD study protocol. BMC Nutr. 2025 Jan 13;11(1):8. doi: 10.1186/s40795-024-00971-6. PMID 39806493